CLINICAL TRIAL: NCT04302883
Title: Transesophageal Echocardiography: Dysphagia Risk in Acute Stroke (T.E.D.R.A.S. Trial)
Acronym: TEDRAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: TEDRAS-1
Record Dates: First submitted 2020-02-19; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Acute Stroke; Dysphagia; Swallowing Disorder
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): TEE FEES
  Interventions: Diagnostic Test: Transesophageal Echocardiography (TEE); Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing
- Control group (Active Comparator): FEES
  Interventions: Diagnostic Test: Transesophageal Echocardiography (TEE); Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography (TEE) — Ultrasound of heart chambers via esophagus
Diagnostic Test: Flexible Endoscopic Evaluation of Swallowing — Endoscopical swallowing study

SUMMARY:
The prevalence of dysphagia in acute stroke patients undergoing transesophageal echocardiography (TEE) is unknown. The aim of this study was to assess for the first time whether TEE has a negative influence on swallowing in acute stroke patients.

DETAILED DESCRIPTION:
Dysphagia is common in patients with acute stroke and deteriorates the overall outcome (1). Transesophageal echocardiography (TEE) is a routine examination in the diagnostic workup of stroke etiology. In cardiac surgery it is known as cause of postoperative dysphagia (2).

Using flexible endoscopic evaluation of swallowing (FEES) T.E.D.R.A.S., as a prospective, blinded, randomized and controlled study, includes patients in two groups in order to test the influence of TEE on swallowing in acute stroke: an intervention group and a control group. FEES is performed for analysis of swallowing in the intervention group (1) one day before TEE, (2) 2-4 hours after TEE, (3) 24 hours after TEE. In the control group FEES is performed on three consecutive days with TEE taking place any time after the last FEES. Validated scores assess dysphagia severity in both groups.

ELIGIBILITY:
Inclusion Criteria:

* acute stroke (max. 7 days post-onset) as displayed by a cranial computed tomography (CT) or magnetic resonance imaging (MRI)
* written informed consent either by patients themselves or by a legal representative
* indication for TEE

Exclusion Criteria:

* brain hemorrhage
* either pre-existing neurogenic dysphagia or
* head-and-neck cancer induced dysphagia
* dementia
* aphasia with an impairment in language comprehension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Secretion severity | Intervention group: One day before TEE; Control group: At least three days before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Murray´s Secretions Severity Rating Scale Minimum value: 0 Maximum value: 3 Higher scores mean worse outcome
Secretion severity | Intervention group: 2-4 hours after TEE; Control group: At least two days before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Murray´s Secretions Severity Rating Scale Minimum value: 0 Maximum value: 3 Higher scores mean worse outcome
Secretion severity | Intervention group: 24 hours after TEE; Control group: At least one day before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Murray´s Secretions Severity Rating Scale Minimum value: 0 Maximum value: 3 Higher scores mean worse outcome
Dysphagia severity | Intervention group: One day before TEE; Control group: At least three days before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Rosenbek´s Penetration-Aspiration-Scale Minimum value: 1 Maximum value: 8 Higher scores mean worse outcome
Dysphagia severity | Intervention group: 2-4 hours after TEE; Control group: At least two days before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Rosenbek´s Penetration-Aspiration-Scale Minimum value: 1 Maximum value: 8 Higher scores mean worse outcome
Dysphagia severity | Intervention group: 24 hours after TEE; Control group: At least one day before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Rosenbek´s Penetration-Aspiration-Scale Minimum value: 1 Maximum value: 8 Higher scores mean worse outcome
Pharyngeal residue severity | Intervention group: One day before TEE; Control group: At least three days before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Yale Pharyngeal Residue Severity Rating Scale Minimum value: 1 Maximum value: 5 Higher scores mean worse outcome
Pharyngeal residue severity | Intervention group: 2-4 hours after TEE; Control group: At least two days before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Yale Pharyngeal Residue Severity Rating Scale Minimum value: 1 Maximum value: 5 Higher scores mean worse outcome
Pharyngeal residue severity | Intervention group: 24 hours after TEE; Control group: At least one day before TEE
  Change in presence and severity of dysphagia examined via FEES and scored by Yale Pharyngeal Residue Severity Rating Scale Minimum value: 1 Maximum value: 5 Higher scores mean worse outcome

SECONDARY OUTCOMES:
Stroke severity | At the day of admission to hospital and up to 2 weeks after TEE
  Quantification of stroke severity via National Institutes of Health Stroke Scale (NIHSS):
  Minimum value: 0 Maximum value: 42 Higher scores mean worse outcome
Degree of disability after stroke | At the day of admission to hospital and up to 2 weeks after TEE
  Measuring the degree of disability or dependance of stroke survivors as measured by the Modified Rankin Scale (MRS):
  Minimum value: 0 Maximum value: 6 Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tibo Gerriets, MD, Principal Investigator — Department of Neurology, University Hospital Giessen
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barer DH. The natural history and functional consequences of dysphagia after hemispheric stroke. J Neurol Neurosurg Psychiatry. 1989 Feb;52(2):236-41. doi: 10.1136/jnnp.52.2.236. PMID 2564884
- [Background] Hogue CW Jr, Lappas GD, Creswell LL, Ferguson TB Jr, Sample M, Pugh D, Balfe D, Cox JL, Lappas DG. Swallowing dysfunction after cardiac operations. Associated adverse outcomes and risk factors including intraoperative transesophageal echocardiography. J Thorac Cardiovasc Surg. 1995 Aug;110(2):517-22. doi: 10.1016/S0022-5223(95)70249-0. PMID 7637370
- [Derived] Hamzic S, Juenemann M, Braun T, Piayda K, Bauer P, Sossalla S, Gerriets T, Khilan H, Butz M, Schramm P, Omar OA. TEDRAS II - transesophageal echocardiography as dysphagia risk in the acute phase of stroke-protocol for a prospective pilot observational trial. Trials. 2025 Oct 27;26(1):445. doi: 10.1186/s13063-025-09065-5. PMID 41146308